CLINICAL TRIAL: NCT02061410
Title: Diagnosis and Treatment of Muscle Inhibition of the Extensor Muscles of the Knee in Elderly
Brief Title: Effects of Neuromuscular Electrical Stimulation (NMES) in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFRGS-2007791
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Knee Osteoarthritis
Keywords: Elderly
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neuromuscular Electrical Stimulation (NMES) (Experimental): The intervention was performed with subjects seated on a regular chair (hip and knee angles maintained at approximately 908), 3 times/week for a period of 8 weeks. NMES parameters included: rectangular biphasic symmetric current, pulse duration of 400 ms and stimulation frequency of 80 Hz.
  Interventions: Device: Neuromuscular Electrical Stimlation (NMES)

INTERVENTIONS:
Device: Neuromuscular Electrical Stimlation (NMES) — The intervention was performed with subjects seated on a regular chair (hip and knee angles maintained at approximately 908), 3 times/week for a period of 8 weeks. NMES parameters included: rectangular biphasic symmetric current, pulse duration of 400 ms and stimulation frequency of 80 Hz.

SUMMARY:
The purpose of this study is to determine the effects of neuromuscular electrical stimulation (NMES) on neuromuscular and functional parameters in elderly with knee osteoarthritis.

The hypothesis is that NAMES is able to strengthen the quadriceps muscle and to improve healthy status of elderly with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* women, minimum age of 50 years;
* clinically diagnosed with knee OA;
* no contraindications to execute maximal knee extension tests (e.g., cardiorespiratory complications);
* no previous musculoskeletal or joint injuries besides knee OA;
* no hip or knee surgery;
* no neurological problems.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Peak torque change | Baseline and 9th intervention week
  Maximal isometric knee extensor torques were obtained on an isokinetic dynamometer (Biodex System 3; Biodex Medical Systems). Participants were positioned on the dynamometer according to the manufacturer's recommendations. After a warm-up and a familiarization session, each subject executed three maximal isometric knee extensor contractions with the knee fixed at a flexion angle of 60o. Each contraction lasted for 5 s and a 2-min interval was observed between consecutive contractions.
Electromyographic activation change | Baseline and 9th intervention week
  An eight channel EMG system (AMT-8, Bortec Biomedical Ltd., Canada) connected to a Windaq data acquisition system (Dataq Instruments Inc., USA) was used during the maximal isometric and concentric knee extensor contractions. EMG signals were obtained following the recommendations by Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles with respect to skin preparation and electrode positioning. Passive bipolar electrodes (Meditrace - 100; Ag/AgCl; inter-electrode distance = 2.2 cm) were placed on the skin covering the rectus femoris, vastus lateralis and vastus medialis muscles. A reference electrode was placed on the medial surface of the tibia. EMG signals were digitized with a sampling frequency of 2000 Hz per channel with a 16 bits analogue-to-digital board DI-720 (Dataq Instruments Inc., USA) and stored for further analysis.
Muscle architecture change | Baseline and 9th intervention week
  An ultrassound system (SSD 4000, 51 Hz, ALOKA Inc., Japan) with a linear array probe (60 mm, 7.5 MHz), was used to determine the thickness, fascicle length, and pennation angle of the vastus lateralis muscle. Ultrassound images were obtained at rest with the subject sitting on the chair of an isokinetic dynamometer (Biodex System 3; Biodex Medical Systems, Shirley, NY) with the hip and knee flexed at 85o and 90o, respectively. All images were captured in the sagittal plane of vastus lateralis (at midway between the lateral condyle of the femur and the greater trochanter). The ultrasound probe was positioned in the approximate direction of the vastus lateralis muscle fibers (long axis with respect to the limb).

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil